CLINICAL TRIAL: NCT02120300
Title: A Phase 2b, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Ledipasvir Fixed-Dose Combination and Sofosbuvir + Ribavirin for Subjects With Chronic Hepatitis C Virus (HCV) and Inherited Bleeding Disorders
Brief Title: Efficacy and Safety of Ledipasvir/Sofosbuvir Fixed-Dose Combination and Sofosbuvir + Ribavirin for Subjects With Chronic Hepatitis C Virus (HCV) and Inherited Bleeding Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-1274
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-10

CONDITIONS: Chronic HCV Infection
MeSH Terms: interventions — ledipasvir, sofosbuvir drug combination; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LDV/SOF GT 1 or 4 (Experimental): Participants with chronic genotypes (GT) 1 or 4 HCV infection will receive LDV/SOF for 12 or 24 weeks. Treatment-experienced cirrhotic participants with genotype 1 HCV infection will receive LDV/SOF for 24 weeks.
  Interventions: Drug: LDV/SOF
- SOF+RBV 12 wks GT 2 (Experimental): Participants with chronic genotype 2 HCV infection will receive SOF+RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- SOF+RBV 24 wks GT 3 (Experimental): Participants with chronic genotype 3 HCV infection will receive SOF+RBV for 24 weeks.
  Interventions: Drug: SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally
  Other Names: Harvoni®; GS-5885/GS-7977
  Arms: LDV/SOF GT 1 or 4
Drug: SOF — 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
  Arms: SOF+RBV 12 wks GT 2; SOF+RBV 24 wks GT 3
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: SOF+RBV 12 wks GT 2; SOF+RBV 24 wks GT 3

SUMMARY:
The primary objectives of this study are to evaluate the antiviral efficacy, safety, and tolerability of treatment with ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) in participants with genotypes 1 and 4 hepatitis C virus (HCV) infection and sofosbuvir (SOF) plus ribavirin (RBV) in participants with genotypes 2 and 3 HCV infection. Participants with an inherited bleeding disorder and chronic HCV infection (either monoinfected or HIV-1/HCV coinfected) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia A, B or C, or Von Willebrand's disease
* Chronic genotype 1, 2, 3 or 4 HCV infection
* HCV RNA ≥ 1000 IU/mL at screening
* Use of protocol specified method(s) of contraception if female of childbearing potential or sexually active male
* Screening laboratory values within defined thresholds
* For HIV-1/HCV co-infected individuals:

  * Suppressed HIV-1 RNA on an antiretroviral (ARV) regimen for at least 6 months prior to screening
  * Stable protocol-approved ARV regimen for > 8 weeks prior to screening
  * CD4 T-cell count > 200 cells/mm^3 at screening

Exclusion Criteria:

* Clinically-significant illness (other than HCV, inherited bleeding disorder or HIV-1) or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol
* Current or prior history of any of the following:

  * Hepatic decompensation
  * Chronic liver disease of a non-HCV etiology
  * Hepatocellular carcinoma (HCC)
  * Infection with hepatitis B virus (HBV)
* Pregnant or nursing female
* Prior treatment with inhibitors of nonstructural protein 5A (NS5A) or the NS5B polymerase
* Chronic use of systemically administered immunosuppressive agents
* For HIV-1/HCV co-infected individuals:

  * Opportunistic infection within 6 months prior to screening
  * Active, serious infection (other than HIV-1 or HCV) requiring parental antibiotics, antivirals or antifungals within 30 days prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Hyland, DPhil, Study Director — Gilead Sciences
Locations (12):
- United States (12):
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Newark, New Jersey
  - New York, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Philadelphia, Pennsylvania

REFERENCES:
- [Background] Walsh C, Workowski K, Terrault N, Sax S, Cohen A, et al. Approved All-Oral Sofosbuvir Regimens Are Safe and Highly Effective in Patients With Hereditary Bleeding Disorders. (2015). Hepatology, 62 (S1): 714A-807A. doi:10.1002/hep.28228

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 10 April 2014. The last study visit occurred on 17 August 2015.
Pre-assignment Details: 147 participants were screened.
Groups:
- LDV/SOF 12 Weeks GT1 or GT4: Ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet once daily for 12 weeks (genotype 1 or 4)
- LDV/SOF 24 Weeks GT1 (TE): LDV/SOF (90/400 mg) FDC tablet once daily for 24 weeks (treatment-experienced [TE] participants with genotype 1 HCV infection and cirrhosis)
- SOF+RBV 12 Weeks GT2: Sofosbuvir (SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 12 weeks (genotype 2)
- SOF+RBV 24 Weeks GT3: SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 24 weeks (genotype 3)
Period: Overall Study
Arm/Group | LDV/SOF 12 Weeks GT1 or GT4 | LDV/SOF 24 Weeks GT1 (TE) | SOF+RBV 12 Weeks GT2 | SOF+RBV 24 Weeks GT3
Started | 101 | 5 | 10 | 6
Completed | 98 | 5 | 10 | 5
Not Completed | 3 | 0 | 0 | 1
Not completed — Enrolled but Never Treated | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LDV/SOF 12 Weeks GT1 or GT4 | LDV/SOF 24 Weeks GT1 (TE) | SOF+RBV 12 Weeks GT2 | SOF+RBV 24 Weeks GT3 | Total
Number analyzed (Participants) | 99 | 5 | 10 | 6 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44 (11.1) | 49 (11.1) | 48 (13.8) | 47 (6.7) | 45 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 1 | 0 | 7
  Male | 93 | 5 | 9 | 6 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 1 | 0 | 5
  Not Hispanic or Latino | 95 | 5 | 9 | 6 | 115
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 18 | 1 | 1 | 0 | 20
  White | 75 | 4 | 8 | 5 | 92
  Asian | 4 | 0 | 1 | 1 | 6
  Other | 2 | 0 | 0 | 0 | 2
Cirrhosis Status [Number; unit: participants]
  No | 71 | 0 | 8 | 4 | 83
  Yes | 28 | 5 | 2 | 2 | 37
HCV Genotype [Number; unit: participants]
  Genotype 1 | 98 | 5 | 0 | 0 | 103
  Genotype 2 | 0 | 0 | 10 | 0 | 10
  Genotype 3 | 0 | 0 | 0 | 6 | 6
  Genotype 4 | 1 | 0 | 0 | 0 | 1
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2 (0.67) | 6.0 (0.85) | 6.2 (1.00) | 6.6 (0.80) | 6.2 (0.71)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 23 | 2 | 2 | 1 | 28
  ≥ 800,000 IU/mL | 76 | 3 | 8 | 5 | 92
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 22 | 2 | 7 | 5 | 36
    CT | 60 | 1 | 3 | 1 | 65
    TT | 17 | 2 | 0 | 0 | 19
HIV Status [Number; unit: participants]
  Negative | 80 | 5 | 6 | 3 | 94
  Positive | 19 | 0 | 4 | 3 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants enrolled into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks GT1 or GT4 | LDV/SOF 24 Weeks GT1 (TE) | SOF+RBV 12 Weeks GT2 | SOF+RBV 24 Weeks GT3
Number analyzed (Participants) | 99 | 5 | 10 | 6
percentage of participants | 99.0 [94.5 to 100.0] | 100.0 [47.8 to 100.0] | 100.0 [69.2 to 100.0] | 83.3 [35.9 to 99.6]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks GT1 or GT4 | LDV/SOF 24 Weeks GT1 (TE) | SOF+RBV 12 Weeks GT2 | SOF+RBV 24 Weeks GT3
Number analyzed (Participants) | 99 | 5 | 10 | 6
percentage of participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks GT1 or GT4 | LDV/SOF 24 Weeks GT1 (TE) | SOF+RBV 12 Weeks GT2 | SOF+RBV 24 Weeks GT3
Number analyzed (Participants) | 99 | 5 | 10 | 6
percentage of participants | 99.0 [94.5 to 100.0] | 100.0 [47.8 to 100.0] | 100.0 [69.2 to 100.0] | 83.3 [35.9 to 99.6]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Weeks 1, 2, 4, 8, 12, 16, 20, and 24
Time Frame: Weeks 1, 2, 4, 8, 12, 16, 20, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks GT1 or GT4 | LDV/SOF 24 Weeks GT1 (TE) | SOF+RBV 12 Weeks GT2 | SOF+RBV 24 Weeks GT3
Number analyzed (Participants) | 99 | 5 | 10 | 6
percentage of participants
  Week 1 | 28.3 | 20.0 | 20.0 | 16.7
  Week 2 | 68.7 | 40.0 | 70.0 | 33.3
  Week 4 | 94.9 | 100.0 | 100.0 | 66.7
  Week 8 | 100.0 | 100.0 | 100.0 | 100.0
  Week 12 | 99.0 | 100.0 | 100.0 | 100.0
  Week 16 | NA — Treatment for this group was only 12 weeks. | 100.0 | NA — Treatment for this group was only 12 weeks. | 100.0
  Week 20 | NA — Treatment for this group was only 12 weeks. | 100.0 | NA — Treatment for this group was only 12 weeks. | 100.0
  Week 24 | NA — Treatment for this group was only 12 weeks. | 100.0 | NA — Treatment for this group was only 12 weeks. | 100.0

5. Secondary Outcome: Change From Baseline in HCV RNA at Weeks 1, 2, 4, 8, 12, 16, 20, and 24
Time Frame: Baseline; Weeks 1, 2, 4, 8, 12, 16, 20, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 12 Weeks GT1 or GT4 | LDV/SOF 24 Weeks GT1 (TE) | SOF+RBV 12 Weeks GT2 | SOF+RBV 24 Weeks GT3
Number analyzed (Participants) | 99 | 5 | 10 | 6
log10 IU/mL
  Baseline | 6.21 (0.673) | 6.02 (0.847) | 6.20 (1.002) | 6.6 (0.803)
  Week 1 (LDV/SOF 12 Weeks: n= 98) | -4.41 (0.580) | -4.32 (0.815) | -4.39 (0.633) | -3.95 (0.473)
  Week 2 (LDV/SOF 24 Week: n=4) | -4.87 (0.642) | -4.65 (0.967) | -5.01 (0.965) | -4.76 (0.797)
  Week 4 | -5.05 (0.662) | -4.87 (0.847) | -5.05 (1.002) | -5.26 (0.786)
  Week 8 | -5.06 (0.673) | -4.87 (0.847) | -5.05 (1.002) | -5.45 (0.803)
  Week 12 (LDV/SOF 12 Weeks: n= 98) | -5.06 (0.675) | -4.87 (0.847) | -5.05 (1.002) | -5.45 (0.803)
  Week 16 | NA (NA) — Treatment for this group was only 12 weeks. | -4.87 (0.847) | NA (NA) — Treatment for this group was only 12 weeks. | -5.45 (0.803)
  Week 20 | NA (NA) — Treatment for this group was only 12 weeks. | -4.87 (0.847) | NA (NA) — Treatment for this group was only 12 weeks. | -5.45 (0.803)
  Week 24 | NA (NA) — Treatment for this group was only 12 weeks. | -4.87 (0.847) | NA (NA) — Treatment for this group was only 12 weeks. | -5.45 (0.803)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks GT1 or GT4 | LDV/SOF 24 Weeks GT1 (TE) | SOF+RBV 12 Weeks GT2 | SOF+RBV 24 Weeks GT3
Number analyzed (Participants) | 99 | 5 | 10 | 6
percentage of participants | 0 | 0 | 0 | 16.7

7. Secondary Outcome: Percentage of Participants That Maintain HIV-1 RNA < 50 Copies/mL at Weeks 4, 8, 12, 16, 20, and 24 (HIV-1/HCV Co-infected Participants Only)
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: Only the participants coinfected with HIV-1 and HCV in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks GT1 or GT4 | SOF+RBV 12 Weeks GT2 | SOF+RBV 24 Weeks GT3
Number analyzed (Participants) | 19 | 4 | 3
percentage of participants
  Week 4 | 100 | 100 | 100
  Week 8 | 100 | 100 | 100
  Week 12 | 100 | 100 | 100
  Week 16 | NA — Treatment for this group was only 12 weeks. | NA — Treatment for this group was only 12 weeks. | 100
  Week 20 | NA — Treatment for this group was only 12 weeks. | NA — Treatment for this group was only 12 weeks. | 100
  Week 24 | NA — Treatment for this group was only 12 weeks. | NA — Treatment for this group was only 12 weeks. | 66.7

8. Secondary Outcome: Change From Baseline in Serum Creatinine at the End of Treatment and at Posttreatment Week 12 (HIV-1/HCV Co-infected Participants Only)
Time Frame: Baseline; Weeks 12, 24, and Posttreatment Week 12
Population: Participants coinfected with HIV-1 and HCV in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | LDV/SOF 12 Weeks GT1 or GT4 | SOF+RBV 12 Weeks GT2 | SOF+RBV 24 Weeks GT3
Number analyzed (Participants) | 19 | 4 | 3
mg/dL
  Baseline | 0.94 (0.197) | 1.01 (0.118) | 0.94 (0.086)
  Week 12 | 0.04 (0.079) | -0.03 (0.095) | -0.03 (0.093)
  Week 24 | NA (NA) — Treatment for this group was only 12 weeks. | NA (NA) — Treatment for this group was only 12 weeks. | -0.08 (0.069)
  Posttreatment Week12 | -0.01 (0.113) | -0.08 (0.015) | -0.02 (0.081)

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | LDV/SOF 12 Weeks GT1 or GT4 | LDV/SOF 24 Weeks GT1 (TE) | SOF+RBV 12 Weeks GT2 | SOF+RBV 24 Weeks GT3
Serious Adverse Events (participants affected / at risk) | 5/99 | 0/5 | 0/10 | 1/6
Other Adverse Events (participants affected / at risk) | 54/99 | 3/5 | 8/10 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks GT1 or GT4 (N=99) | LDV/SOF 24 Weeks GT1 (TE) (N=5) | SOF+RBV 12 Weeks GT2 (N=10) | SOF+RBV 24 Weeks GT3 (N=6)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Miscarriage of partner (Social circumstances) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks GT1 or GT4 (N=99) | LDV/SOF 24 Weeks GT1 (TE) (N=5) | SOF+RBV 12 Weeks GT2 (N=10) | SOF+RBV 24 Weeks GT3 (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 29 | 1 | 3 | 2
Influenza like illness (General disorders) | 1 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 8 | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
Osteorrhagia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 6 | 0 | 1 | 0
Headache (Nervous system disorders) | 14 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 5 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 6 | 0 | 1 | 3
Irritability (Psychiatric disorders) | 2 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years